CLINICAL TRIAL: NCT01572675
Title: Pharmacoepidemiological Study on the Use of Arcoxia® Under Actual Conditions of Use in France
Brief Title: A Study of the Patterns of Use of Etoricoxib in France (MK-0663-148)
Acronym: COXIBUS
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0663-148
Record Dates: First submitted 2012-02-03; First posted 2012-04-06 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Pharmacoepidemiological; Longitudinal; Observational
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib; Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group Arcoxia®: Participants who were either previously treated with Arcoxia® or initiated on study treatment with Arcoxia®. Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
  Interventions: Drug: etorocoxib
- Group Celebrex®: Participants who were either previously treated with Celebrex® or initiated on study treatment with Celebrex®. Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: etorocoxib — Administered as 30 mg or 60 mg oral film-coated tablets
  Other Names: Arcoxia®
  Groups: Group Arcoxia®
Drug: celecoxib — Administered as 100 mg or 200 mg oral hard capsules
  Other Names: Celebrex®
  Groups: Group Celebrex®

SUMMARY:
This postmarketing study will examine the use of etoricoxib (Arcoxia®) in routine clinical practice in France as well as the use of celecoxib (Celebrex®).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive, discontinued the previous treatment course of etoricoxib or celecoxib at least 3 months previously or currently receiving continuous treatment with oral etoricoxib or celecoxib
* Consent to take part in the study
* Included in his/her physician's client base for at least 1 year

Exclusion Criteria:

* Unable to receive follow-up over a year
* Included in an interventional trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants spontaneously consulting a general practitioner or rheumatologist and having agreed to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 621 total participants were screened; 71 participants were excluded for inclusion criteria violation and 3 were excluded for unavailability of informed consent.
Period: Overall Study
Arm/Group | Group Arcoxia® | Group Celebrex®
Started | 268 | 279
Completed | 31 | 56
Not Completed | 237 | 223
Not completed — End of prescribed treatment | 140 | 118
Not completed — Recovery | 16 | 23
Not completed — Lack of Efficacy | 31 | 31
Not completed — Intolerance | 6 | 5
Not completed — Improved symptoms | 8 | 2
Not completed — Surgical intervention | 3 | 6
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Death unrelated to coxibs | 1 | 1
Not completed — Other disease detected | 1 | 1
Not completed — Unknown reason | 1 | 1
Not completed — Rheumatologist new evaluation | 0 | 1
Not completed — Missing data | 1 | 4
Not completed — Lost to Follow-up | 22 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Arcoxia® | Group Celebrex® | Total
Number analyzed (Participants) | 268 | 279 | 547
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (13.8) | 62.4 (14.2) | 61.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 179 | 345
  Male | 102 | 100 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Proper Use of Arcoxia® and Celebrex®
Description: Proper use of study medication is defined as administration of medication in terms of indication and dosage according to Market Authorization (MA). Proper use of Arcoxia® is defined as administration of a starting dose of 30 mg daily, not to exceed 60 mg daily during follow-up, for the treatment of symptoms of osteoarthritis. Proper use of Celebrex® is defined as administration of a starting dose of 200 mg daily, not to exceed 400 mg daily during follow-up, for easing symptoms in the treatment of osteoarthritis, rheumatoid arthritis, and ankylosing spondylitis. Data to assess proper use were collected through use of a medical questionnaire and patient form. Data pertaining to indication was collected by open-field to allow physicians to precisely indicate the reason for prescription. Recorded indications were then analyzed by two medical experts (an independent expert and a member of the Scientific Community) to assess proper use or misuse.
Time Frame: Up to 12 months
Population: All participants with complete data relative to correct use of the coxib and at least 1 data point relative to misuse of the coxib.
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 257 | 264
Participants | 65 | 118

2. Primary Outcome: Reasons for Misuse of Arcoxia® and Celebrex®
Description: Proper use of study medication is defined as administration of medication in terms of indication and dosage according to MA. Proper use of Arcoxia® is defined as administration of a starting dose of 30 mg daily, not to exceed 60 mg daily during follow-up, for the treatment of symptoms of osteoarthritis. Proper use of Celebrex® is defined as administration of a starting dose of 200 mg daily, not to exceed 400 mg daily during follow-up, for easing symptoms in the treatment of osteoarthritis, rheumatoid arthritis, and ankylosing spondylitis. Data to assess proper use were collected through use of a medical questionnaire and patient form. Data pertaining to indication was collected by open-field to allow physicians to precisely indicate the reason for prescription. Recorded indications were then analyzed by two medical experts (an independent expert and a member of the Scientific Community) to assess proper use or misuse.
Time Frame: Up to 12 months
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (misuse)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 192 | 146
Participants
  Non-MA-Compliant Indication | 83 | 114
  Non-MA-Compliant Starting Dose | 62 | 19
  Non-MA-Compliant Starting Dose and Indication | 46 | 13
  Non-MA-Compliant Indication & Dose (Starting &Max) | 1 | 0

3. Primary Outcome: Indications for Which Arcoxia® and Celebrex® Were Prescribed
Description: The reasons (indications) for prescribing of Arcoxia® or Celebrex® were collected in open-field forms by the Investigator; category assignment (i.e, re-codification) of verbatim entries was conducted by a group of medical experts under the guidance approved by the MA. This endpoint gives the number of participants treated per indication.
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (indication)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 264 | 275
Participants
  Other pain (e.g., spinal pain, joint pain) | 113 | 117
  Osteoarthritis | 105 | 104
  Inflammatory rheumatism | 13 | 18
  Neuralgia | 17 | 24
  Non-joint rheumatism | 12 | 12
  Unclassified arthropathy | 4 | 0
  Missing data | 4 | 4

4. Primary Outcome: Dosage of Arcoxia® and Celebrex® at Initiation
Description: Dosage at initiation of treatment with Arcoxia® or Celebrex® was identified. MA compliant dosage at initiation corresponds to a (starting) dose of 30 mg daily for Arcoxia® or a (starting) dose of 200 mg daily for Celebrex®. The dose for initiation was calculated by multiplying the number of doses per day with the dose level (total daily dose) as noted in the prescription record.
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (dosage at initiation)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 268 | 279
Participants
  30 mg | 151 | 0
  60 mg | 107 | 0
  > 60 mg; <100 mg | 1 | 0
  100 mg | 0 | 23
  >100 mg; < 200 mg | 1 | 0
  200 mg | 0 | 219
  400 mg | 0 | 32
  > 400 mg | 0 | 0

5. Primary Outcome: Mean Dosage of Arcoxia® and Celebrex® During Treatment
Description: The mean dosage of Arcoxia® and Celebrex® during treatment was determined. For participants who stopped treatment after their initial study visit, the maximum dose recorded at their final study visit was considered when calculating their mean dosage during treatment.
Time Frame: Up to 12 months
Population: All participants who discontinued treatment during follow-up or were still on treatment after one year of follow-up under protocol; participants who were lost to follow-up were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 246 | 252
mg/day | 44.1 (14.8) | 221.9 (73.1)

6. Primary Outcome: Number of Participants Requiring Dose Modification of Arcoxia® and Celebrex®
Description: Participants requiring modifications to their Arcoxia® or Celebrex® dose regimens during their on study treatment course were identified. Dose modifications were defined as an increase, decrease followed by increase, decrease, or increase followed by decrease in the participant's daily dose; all categorizations were exclusive. If the maximum dose at discontinuation of treatment was greater than that at initiation, the participant was considered as having had an increase in dose during treatment. Alternatively, if data obtained from a participant's prescription records showed a successive lowering of dosage, the participant was considered as having had a decrease in dose during treatment. Dosages at baseline were included in the dose modification determination for treatment renewal participants.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 246 | 252
Participants
  Missing data | 1 | 5
  Dose increase | 42 | 33
  Dose decrease followed by increase | 1 | 0
  Dose decrease | 2 | 5
  Dose increase followed by decrease | 0 | 3

7. Primary Outcome: Duration of Prescription for Arcoxia® and Celebrex® at Enrollment
Description: The mean duration of prescription at enrollment for participants treated with Arcoxia® and Celebrex® was determined using the participant's record.
Time Frame: Up to 3 months prior to study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (duration of prescription)
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Group Arcoxia® - Initiation: Participants who initiated on study treatment with Arcoxia® (treatment-naïve or had discontinued treatment at least 3 months prior). Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
- Group Arcoxia® - Renewal: Participants who started Arcoxia® prior to study entry (prescription renewal). Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
- Group Celebrex® - Initiation: Participants who initiated on study treatment with Celebrex® (treatment-naïve or had discontinued treatment at least 3 months prior). Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
- Group Celebrex® - Renewal: Participants who started Celebrex® prior to study entry (prescription renewal). Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 119 | 157 | 268 | 276
Days | 25.5 (18.4) | 38.1 (24.1) | 23.9 (17.6) | 41.7 (26.9) | 31.1 (22.0) | 34.0 (24.9)
Statistical Analysis 1: Comparison: Group Arcoxia® - Initiation vs Group Arcoxia® - Renewal; Group comparison (Arcoxia® [Initiation] vs Arcoxia® [Renewal]) for duration of prescription at enrollment; Test type: Superiority or Other; p < 0.001, p-student
Statistical Analysis 2: Comparison: Group Celebrex® - Initiation vs Group Celebrex® - Renewal; Group comparison (Celebrex® [Initiation] vs Celebrex® [Renewal]) for duration of prescription at enrollment; Test type: Superiority or Other; p < 0.001, p-student

8. Primary Outcome: Total Duration of Treatment With Arcoxia® and Celebrex®
Description: The total duration of treatment (DoT) with Arcoxia® or Celebrex® was determined for populations that achieved end-of study and end-of-protocol or that were categorized as lost to follow-up. Participants enumerated as end-of-study had their treatment discontinued during the protocol-specified one year of follow-up. Participants enumerated as end-of-protocol were ongoing treatment at end of the protocol-specified one year of follow-up. Participants categorized as lost to follow-up had no follow-up visit where a determination of discontinuation from treatment could be made.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 251 | 256
Days
  DoT - End-of-study participants (n=215,196) | 85.2 (127.1) | 117.8 (307.6)
  DoT - End-of-protocol participants (n=31,56) | 472.9 (90.7) | 595.2 (456.7)
  DoT - Lost to follow-up participants (n=5,4) | 122.4 (131.6) | 142.0 (128.8)

9. Primary Outcome: Maximum Dosage Prescribed During Treatment With Arcoxia® and Celebrex®
Description: Mean maximum dosage prescribed during follow-up in participants treated with Arcoxia® or Celebrex®. Dosage is expressed as total daily dose.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 137 | 109 | 109 | 143 | 246 | 252
mg/day | 47.1 (16.2) | 48.4 (14.7) | 228.4 (79.5) | 242.7 (86.0) | 47.7 (15.5) | 236.5 (83.4)

10. Primary Outcome: Reasons for Discontinuation of Treatment With Arcoxia® and Celebrex®
Description: The individual reasons for discontinuation of treatment with Arcoxia® or Celebrex® were identified over the course of study through either physician selection from a pre-determined list or verbatim entry by the physician with subsequent re-codification by Sponsor.
Time Frame: Up to 12 months
Population: All participants who discontinued treatment during follow-up under protocol; participants who were lost to follow-up were excluded from this analysis.
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 215 | 196
Participants
  End of prescribed treatment | 140 | 118
  Recovery | 16 | 23
  Lack of efficacy | 31 | 31
  Intolerance | 6 | 5
  Improved symptoms | 8 | 2
  Surgical intervention | 3 | 6
  Participant decision | 5 | 1
  Physician decision | 2 | 2
  Death unrelated to coxibs | 1 | 1
  Other disease detected | 1 | 1
  Other - unknown reason | 1 | 1
  Rheumatologist new evaluation | 0 | 1
  Missing data | 1 | 4

11. Primary Outcome: Type of Arcoxia® and Celebrex® Use
Description: The type of Arcoxia® or Celebrex® use during the study was classified as continuous (without interruption >7 days) or intermittent (with interruption >7 days) by the Investigating Physician at time of treatment discontinuation.
Time Frame: Up to 12 months
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 215 | 194
Participants
  Missing data | 0 | 2
  Intermittent | 44 | 47
  Continuous | 171 | 147

12. Primary Outcome: Type of Arcoxia® and Celebrex® Use According to Duration of Treatment
Description: Use of selective cyclooxygenase-2 (COX-2) inhibitors (Arcoxia® and Celebrex®) as assessed by the Investigating Physician at time of treatment discontinuation was correlated to the overall duration of treatment experienced by the participant (i.e., intermittent or continuous selective COX-2 inhibitor use vs. total participant time on treatment). Type of use was classified as continuous (without interruption >7 days) or intermittent (with interruption >7 days). Four successive treatment intervals were assessed in this endpoint: 1) Up to thirty days of treatment 2) From one to three months of treatment 3) From three months to one year of treatment and 4) More than one year of treatment.
Time Frame: Up to 12 months
Population: as for outcome 10
Measure: Number; unit: Participants
Groups:
- Up to Thirty Days: Participants who were either previously treated with Arcoxia® or Celebrex® or initiated on study treatment with Arcoxia® or Celebrex® and were treated for ≤ 30 days
- From One to Three Months: Participants who were either previously treated with Arcoxia® or Celebrex® or initiated on study treatment with Arcoxia® or Celebrex® and were treated from one to three months total
- From Three Months to One Year: Participants who were either previously treated with Arcoxia® or Celebrex® or initiated on study treatment with Arcoxia® or Celebrex® and were treated from three months to one year
- More Than One Year: Participants who were either previously treated with Arcoxia® or Celebrex® or initiated on study treatment with Arcoxia® or Celebrex® and were treated for more than one year
Arm/Group | Up to Thirty Days | From One to Three Months | From Three Months to One Year | More Than One Year
Number analyzed (Participants) | 206 | 112 | 75 | 18
Participants
  Missing data | 0 (127.1) | 1 (307.6) | 1 | 0
  Intermittent | 24 (90.7) | 38 (456.7) | 22 | 7
  Continuous | 182 (131.6) | 73 (128.8) | 52 | 11
Statistical Analysis 1: Comparison: Up to Thirty Days vs More Than One Year; Duration of treatment comparison (More than one year vs Up to thirty days) for intermittent selective COX-2 inhibitor use. The analysis assessed whether long-term treatment was more correlated with intermittent selective COX-2 inhibitor use compared to short-term treatment; Test type: Superiority or Other; p < 0.001, Chi-squared

13. Secondary Outcome: Mean Body Mass Index (BMI) at Study Entry in Participants Treated With Arcoxia® and Celebrex®
Description: Participants' BMI was assessed at study entry by the Investigating Physician. BMI is calculated as the participant's weight in kilograms (kg) divided by height in meters squared. BMI under 18.5 is commonly considered underweight; within the range (18.5 to 25) as normal weight; within the range (25 to 30) as overweight; and over 30 as obese.
Time Frame: At study entry (baseline)
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (BMI)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 147 | 119 | 120 | 158 | 266 | 278
kg/m^2 | 26.6 (5.2) | 27.1 (4.5) | 27.3 (4.5) | 27.0 (5.6) | 26.8 (4.9) | 27.1 (5.1)

14. Secondary Outcome: Mean Systolic and Diastolic Blood Pressure (BP) at Study Entry in Participants Treated With Arcoxia® and Celebrex®
Description: Mean systolic blood pressure (SBP) and diastolic blood pressure (DBP) were assessed at study entry by the Investigating Physician. Definition of controlled BP: SBP <140 mmHg and DBP <90 mmHg. Definition of uncontrolled BP: SBP ≥140 mmHg and/or DBP ≥90 mmHg.
Time Frame: At study entry (baseline)
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (SBP and DBP)
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 146 | 118 | 116 | 158 | 264 | 274
mmHG
  SBP | 127.4 (10.7) | 130.9 (9.9) | 127.9 (9.5) | 128.4 (8.2) | 129.0 (10.4) | 128.2 (8.8)
  DBP | 76.0 (7.0) | 76.8 (7.3) | 76.0 (7.6) | 75.1 (7.1) | 76.4 (7.1) | 75.4 (7.3)

15. Secondary Outcome: Blood Pressure at Study Entry in Participants Treated With Arcoxia® and Celebrex®
Description: Participants' BP (SBP/DBP) was assessed at study entry by the Investigating Physician. Definition of controlled BP: SBP <140 mmHg and DBP <90 mmHg. Definition of uncontrolled BP: SBP ≥140 mmHg and/or DBP ≥90 mmHg.
Time Frame: At study entry (baseline)
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (BP)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  MIssing data | 3 (10.7) | 1 (9.9) | 5 (9.5) | 0 (8.2) | 4 (10.4) | 5 (8.8)
  <120/80 mmHg | 15 (7.0) | 5 (7.3) | 8 (7.6) | 6 (7.1) | 20 (7.1) | 14 (7.3)
  120 mmHg ≤SBP<140 mmHg and/or 80 mmHg ≤DBP<90 mmHg | 105 | 80 | 87 | 127 | 185 | 214
  140 mmHg ≤SBP<180 mmHg and/or 90 mmHg≤DBP<100 mmHg | 26 | 33 | 21 | 25 | 59 | 46
  SBP≥180 mmHg and/or DBP≥110 mmHg | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group Arcoxia® vs Group Celebrex®; Group comparison (Arcoxia® vs Celebrex®) for controlled BP (SBP <140 mmHg and DBP <90 mmHg) at study entry; Test type: Superiority or Other; p = 0.104, Chi-squared
Statistical Analysis 2: Comparison: Group Arcoxia® - Initiation vs Group Arcoxia® - Renewal; Group comparison (Arcoxia® [Initiation] vs Arcoxia® [Renewal]) for controlled BP (SBP <140 mmHg and DBP <90 mmHg) at study entry; Test type: Superiority or Other; p = 0.0049, Chi-squared
Statistical Analysis 3: Comparison: Group Celebrex® - Initiation vs Group Celebrex® - Renewal; Group comparison (Celebrex® [Initiation] vs Celebrex® [Renewal]) for controlled BP (SBP <140 mmHg and DBP <90 mmHg) at study entry; Test type: Superiority or Other; p = 0.618, Chi-squared

16. Secondary Outcome: Medical History of Participants Treated With Arcoxia® and Celebrex®
Description: Relevant medical history of participants treated with Arcoxia® or Celebrex® was recorded by the Investigating Physician.
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (medical history)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  Arterial hypertension (n=146,118,116,156,264,272) | 37 | 47 | 34 | 58 | 84 | 92
  Acute rhinitis (n=145,115,115,157,260,272) | 20 | 15 | 10 | 12 | 35 | 22
  Bronchospam (n=145,117,115,158,262,273) | 9 | 6 | 2 | 6 | 15 | 8
  Urticaria (n=146,116,115,156,262,271) | 5 | 5 | 0 | 4 | 10 | 4
  Peptic ulcer/bleeding (n=146,118,117,158,264,275) | 5 | 0 | 3 | 4 | 5 | 7
  Angioedema (n=145,117,114,157,262,271) | 2 | 0 | 1 | 2 | 2 | 3
  Nasal polyps (n=146,116,114,158,262,272) | 0 | 1 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Group Arcoxia® - Initiation vs Group Arcoxia® - Renewal; Group comparison (Arcoxia® [Initiation] vs Arcoxia® [Renewal]) for medical history of arterial hypertension; Test type: Superiority or Other; p = 0.012, Chi-squared
Statistical Analysis 2: Comparison: Group Celebrex® - Initiation vs Group Celebrex® - Renewal; Group comparison (Celebrex® [Initiation] vs Celebrex® [Renewal]) for medical history of arterial hypertension; Test type: Superiority or Other; p = 0.175, Chi-squared

17. Secondary Outcome: Co-morbidities in Participants Treated With Arcoxia® and Celebrex®
Description: Associated co-morbidities at study entry (baseline) in participants treated with Arcoxia® or Celebrex® were recorded by the Investigating Physician. CHF/IHD/PAD = Congestive heart failure/Ischemic heart disease/Peripheral artery disease
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (co-morbidities)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  At least one co-morbidity | 55 | 44 | 32 | 62 | 99 | 94
  Hyperlipidemia | 43 | 34 | 26 | 46 | 77 | 72
  Diabetes | 14 | 11 | 6 | 22 | 25 | 28
  Hepatic insufficiency | 4 | 3 | 0 | 2 | 7 | 2
  Inflammatory bowel disease | 2 | 4 | 3 | 1 | 6 | 4
  CHF/IHD/PAD | 1 | 2 | 3 | 6 | 3 | 9
  Active peptic ulceration/ GI bleeding | 1 | 0 | 0 | 0 | 1 | 0
  Missing data | 5 | 2 | 4 | 0 | 7 | 4

18. Secondary Outcome: Significant Past Treatments Prior to Initiating Treatment With Arcoxia® or Celebrex®
Description: 'Significant' treatments that preceded the use of selective COX-2 inhibitors (Arcoxia® or Celebrex®) were identified using a closed-ended (yes/ no/ do not know) questionnaire. Significant is defined as associated with a chronic disease or having a potential link with participant's current use of a selective COX-2 inhibitors (Arcoxia® or Celebrex®). ARBs = Angiotensin 2 receptor blockers. ACEIs = Angiotensin-converting enzyme inhibitors. SSRIs = Selective serotonin reuptake Inhibitors. PAIs = Platelet aggregation inhibitors.
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (past treatments)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  At least one treatment (n=146,118,117,158,264,275) | 102 | 75 | 67 | 118 | 177 | 185
  Proton-pump inhibitors (n=146,115,116,156,261,272) | 58 | 43 | 30 | 65 | 101 | 95
  Hypolipidemic agents (n=146,116,117,156,262,273) | 39 | 32 | 24 | 45 | 71 | 69
  ARBs (n=144,115,116,155,259,271) | 22 | 29 | 23 | 37 | 51 | 60
  Diuretics (N=146,117,117,156,263,273) | 16 | 24 | 10 | 29 | 40 | 39
  ACEIs (n=145,116,117,157,261,274) | 11 | 22 | 13 | 20 | 33 | 33
  SSRIs (n=146,116,117,158,262,275) | 15 | 15 | 8 | 25 | 30 | 33
  Anti-diabetic agents (n=146,115,117,158,261,275) | 14 | 8 | 6 | 19 | 22 | 25
  Histamine H2 blockers (n=146,117,117,156,263,273) | 14 | 14 | 7 | 20 | 28 | 27
  PAIs (n=146,118,117,158,264,275) | 5 | 8 | 6 | 8 | 13 | 14
  Oral anticoagulants (n=146,118,117,158,264,275) | 1 | 4 | 3 | 6 | 5 | 9
  Alpha-blockers (n=146,116,117,157,262,274) | 1 | 1 | 4 | 5 | 2 | 9
Statistical Analysis 1: Comparison: Group Arcoxia® - Initiation vs Group Arcoxia® - Renewal; Group comparison (Arcoxia® [Initiation] vs Arcoxia® [Renewal]) for significant past treatments; Test type: Superiority or Other; p = 0.701, Chi-squared
Statistical Analysis 2: Comparison: Group Celebrex® - Initiation vs Group Celebrex® - Renewal; Group comparison (Celebrex® [Initiation] vs Celebrex® [Renewal]) for significant past treatments; Test type: Superiority or Other; p = 0.007, Chi-squared
Statistical Analysis 3: Comparison: Group Arcoxia® vs Group Celebrex®; Group comparison (Arcoxia® vs Celebrex®) for significant past treatments; Test type: Superiority or Other; p = 0.955, Chi-squared

19. Secondary Outcome: Medications Co-Prescribed at Study Entry in Participants Treated With Arcoxia® and Celebrex®
Description: Concomitant medications prescribed to participants treated with Arcoxia® and Celebrex® were collected via the physician prescription note at time of participant's study entry. NSAIDS = Non-steroidal anti-inflammatory agents.
Time Frame: At study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (co-prescriptions at entry)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  Missing data | 15 | 22 | 3 | 23 | 37 | 26
  At least one treatment | 95 | 89 | 73 | 120 | 184 | 193
  Analgesics | 52 | 66 | 38 | 75 | 118 | 113
  Cardiovascular agents | 30 | 40 | 31 | 59 | 70 | 90
  Digestive system agents | 37 | 33 | 22 | 61 | 70 | 83
  Nervous system agents | 17 | 24 | 14 | 45 | 41 | 59
  NSAIDS | 25 | 21 | 15 | 28 | 46 | 43
  Rheumatologic agents | 17 | 21 | 23 | 29 | 38 | 52
  Metabolic system agents | 14 | 23 | 11 | 38 | 37 | 49
  Respiratory system agents | 9 | 16 | 7 | 21 | 25 | 28
  Hormonal agents | 8 | 13 | 6 | 15 | 21 | 21
  Hematologic agents | 1 | 10 | 6 | 16 | 11 | 22
  Urinary-genital system agents | 4 | 4 | 6 | 12 | 8 | 18
  Dermatological agents | 7 | 1 | 4 | 14 | 8 | 18
  Anti-infectious agents | 4 | 4 | 2 | 12 | 8 | 14
  Other not-classified | 6 | 5 | 5 | 23 | 11 | 28

20. Secondary Outcome: Medications Co-Prescribed Over the Course of Follow-up With Arcoxia® and Celebrex®
Description: Concomitant medications prescribed during the course of follow-up to participants treated with Arcoxia® and Celebrex® were extracted from participants' medical records. NSAIDS = Non-steroidal anti-inflammatory agents.
Time Frame: Up to 12 months
Population: All participants in compliance with study inclusion criteria with at least one follow-up visit (with an available prescription file) other than the end-of-study visit were used for analysis of the endpoint
Measure: Number; unit: Participants
Groups:
- Group Arcoxia®: Participants who either previously received Arcoxia® or initiated on study treatment with Arcoxia®. Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
- Group Celebrex®: Participants who either previously received Celebrex® or initiated on study treatment with Celebrex®. Participant data in terms of dosage, treatment duration, and reasons for prescription was collected under actual conditions of use.
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 104 | 116
Participants
  Missing data | 26 | 38
  At least one treatment | 75 | 65
  Analgesics | 58 | 55
  Cardiovascular agents | 41 | 39
  Digestive system agents | 39 | 36
  Nervous system agents | 25 | 32
  Respiratory system agents | 32 | 23
  Metabolic system agents | 28 | 22
  Rheumatologic agents | 19 | 20
  NSAIDS | 17 | 21
  Anti-infectious agents | 16 | 16
  Hormonal agents | 12 | 13
  Dermatological agents | 13 | 12
  Hematologic agents | 14 | 8
  Urinary-genital system agents | 8 | 8
  Other | 17 | 17

21. Secondary Outcome: Number of Participants Treated With Other Agents Prior to Initiation of Arcoxia® and Celebrex®
Description: Other prescribed agents for the same study indication within 3 months preceding the decision to initiate treatment with selective COX-2 inhibitors (Arcoxia® or Celebrex®) were determined using the participant's medical record. NSAIDS = Non-steroidal inflammatory agents.
Time Frame: Up to 3 months prior to study entry
Population: The per protocol analysis population consisting of all participants in compliance with study inclusion criteria with data of sufficient quality for analysis of the endpoint (other prior agents)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Celebrex® - Initiation | Group Celebrex® - Renewal | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 149 | 119 | 121 | 158 | 268 | 279
Participants
  At least one treatment (n=146,118,117,158,264,275) | 93 | 86 | 62 | 102 | 179 | 164
  Paracetamol (n=146,118,117,158,264,275) | 83 | 82 | 54 | 90 | 165 | 144
  NSAIDS (n=146,118,117,158,264,275) | 33 | 19 | 19 | 23 | 52 | 42
  Analgesics (n=146,118,117,158,264,275) | 4 | 4 | 1 | 7 | 8 | 8
  Corticosteroids (n=140,107,111,152,247,263) | 7 | 3 | 6 | 13 | 10 | 19
Statistical Analysis 1: Comparison: Group Arcoxia® vs Group Celebrex®; Group comparsion (Arcoxia® vs Celebrex®) for previous treatment with other agents prior to initiation of Arcoxia® and Celebrex® for the main study indications; Test type: Superiority or Other; p = 0.049, Fisher Exact

22. Secondary Outcome: Number of Participants Switching to Another Treatment With the Same Reason for Prescription
Description: Participants who switched to another NSAID or other therapy for the same reason for prescription upon discontinuation of treatment with Arcoxia® or Celebrex® were determined.
Time Frame: Up to 12 months
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 215 | 196
Participants
  Prescription of a new treatment | 33 | 29
  NSAIDS | 22 | 22
  Analgesics | 9 | 6
  Other (TNF-alpha inhibitors, corticosteroids) | 1 | 1

23. Secondary Outcome: Number of Participants With Contraindications for Use of Arcoxia®
Description: Participants noted with contraindications for use of Arcoxia® according to the MA during initiation of treatment are described. CHF = congestive heart failure. HA = hepatic impairment. IBD = inflammatory bowel disease. IHD = ischemic heart disease. PAD = peripheral artery disease.
Time Frame: At study entry
Population: The safety population consisting of all participants who enrolled in the study with data of sufficient quality for analysis of the endpoint (contraindications)
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® - Initiation | Group Arcoxia® - Renewal | Group Arcoxia®
Number analyzed (Participants) | 149 | 119 | 268
Participants
  At least one contraindication (n=122,100,122) | 36 | 34 | 70
  One total contraindication (n=36,34,70) | 29 | 32 | 61
  Two total contraindications (n=36,34,70) | 7 | 2 | 9
  History of acute rhinitis (n=145,115,260) | 20 | 15 | 35
  Creatinine clearance <30 ml/min (n=125,108,233) | 1 | 0 | 1
  History of bronchospasm (n=145,117,262) | 9 | 6 | 15
  History of urticaria (n=146,116,262) | 5 | 5 | 10
  Presence of IBD (n=146,118,264) | 2 | 4 | 6
  Presence of CHF (n=146,118,264) | 0 | 2 | 2
  Presence of IHD and/or PAD (n=142,118,260) | 1 | 2 | 3
  History of allergic reaction (n=145,118,263) | 1 | 0 | 1
  History of nasal polyps (n=146,116,262) | 0 | 1 | 1
  Blood pressure not controlled (n=146,118,264) | 1 | 0 | 1
  History of angioedema (n=145,117,262) | 2 | 0 | 2
  Patients with severe HA (n=146,118,264) | 1 | 0 | 1
  <16 years of age (n=149,119,268) | 0 | 0 | 0
  Pregnancy or lactation (n=92,73,165) | 0 | 1 | 1

24. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to 12 months
Population: The safety population consisting of all participants who enrolled in the study
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 268 | 279
Participants | 10 | 5
Statistical Analysis 1: Comparison: Group Arcoxia® vs Group Celebrex®; Group comparsion (Arcoxia® vs Celebrex®) of adverse events experienced during treatment; Test type: Superiority or Other; p = 0.165, Chi-squared

25. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: Discontinuation/withdrawal of study treatment due to an adverse event was performed at the discretion of the investigator or the Sponsor for safety concerns. An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
Time Frame: Up to 12 months
Population: The safety population consisting of all participants who enrolled in the study
Measure: Number; unit: Participants
Arm/Group | Group Arcoxia® | Group Celebrex®
Number analyzed (Participants) | 268 | 279
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All participants who enrolled in the study were included in the safety reporting.
Arm/Group | Group Arcoxia® | Group Celebrex®
Serious Adverse Events (participants affected / at risk) | 0/268 | 0/279
Other Adverse Events (participants affected / at risk) | 0/268 | 0/279

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No